CLINICAL TRIAL: NCT04701008
Title: Observational Study of the Efficacy of Ketamine for Rescue Analgesia in the Post Anesthesia Recovery Room
Brief Title: Efficacy of Ketamine in Post Anesthesia Recovery Room
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00102967
Record Dates: First submitted 2021-01-05; First posted 2021-01-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-07

CONDITIONS: Pain, Postoperative; Ketamine Adverse Reaction; Pain, Refractory; Pain, Intractable; Pain, Acute
Keywords: pain score reduction; reduction in pain scores; post-operative pain; ketamine use in recovery room; recovery room; ketamine recovery; ketamine rescue
MeSH Terms: conditions — Pain, Postoperative; Pain, Intractable; Acute Pain | interventions — Ketamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with significative post-operative pain despite: Patients with significant pain despite receiving narcotics in PACU will receive a bolus dose of IV ketamine to assess its efficacy for pain score reduction. Bolus doses are given by 10mg IV increments, to reach approximate dose of 0,25mg/kg.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — IV ketamine - 10mg bolus may be repeated repeated 2-3 times depending on clinical judgement

SUMMARY:
Observational study to assess efficacy of IV ketamine bolus when used in the post anesthesia recovery unit for uncontrolled pain despite use of opioids.

DETAILED DESCRIPTION:
In this observational study, the investigators will monitor all patients with significant pain after any non-cardiac surgical intervention at the University of Alberta Hospital.

After receiving an adequate dose of potent opioids (hydromorphone, morphine), the participants will receive up to 0,2-0,25 mg/kg IV ketamine bolus. In our center these boluses are given with 10-20mg increments.

The adequate dose of opioids will be determined by the attending anesthesiologist, depending on what patients received intraoperatively and on their comorbidities.

Pain scores will be assessed before and after administration of this drug. The incidence of any side effect after ketamine administration will be documented.

ELIGIBILITY:
Inclusion Criteria:

Adult patients undergoing non cardiac surgery at University of Alberta Hospital meeting the following criteria:

* age ≥ 18
* significant pain despite narcotics used in post-anesthesia care unit
* ketamine ordered by attending anesthesiologist

Exclusion Criteria:

* Patient refusal to receive ketamine
* Patients undergoing cardiac surgery
* Patients who received no narcotics
* Contra-indication to receiving ketamine (determined by attending anesthesiologist)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The following patients will be identified and recruited at the post-anesthesia care unit:
  Adult patients undergoing non-cardiac surgery at University of Alberta Hospital meeting the following criteria:
  1. age ≥ 18
  2. significant pain despite narcotics used in post anesthesia care unit
  3. ketamine ordered by attending anesthesiologist
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Reduction in pain score after ketamine use in PACU | in the immediate post-operative period in recovery room
  The Numeric Rating Scale (NRS-11) is an 11-point scale for patient self-reporting of pain. It is what is used most often in our recovery room for pain assessment. A score of 0/10 means no pain, and 10/10 means worst pain.

SECONDARY OUTCOMES:
Incidence of side effects after ketamine use | in the immediate post-operative period in recovery room

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brinck EC, Tiippana E, Heesen M, Bell RF, Straube S, Moore RA, Kontinen V. Perioperative intravenous ketamine for acute postoperative pain in adults. Cochrane Database Syst Rev. 2018 Dec 20;12(12):CD012033. doi: 10.1002/14651858.CD012033.pub4. PMID 30570761
- [Background] Gillies A, Lindholm D, Angliss M, Orr A. The use of ketamine as rescue analgesia in the recovery room following morphine administration--a double-blind randomised controlled trial in postoperative patients. Anaesth Intensive Care. 2007 Apr;35(2):199-203. PMID 17444308
- [Background] Weinbroum AA. A single small dose of postoperative ketamine provides rapid and sustained improvement in morphine analgesia in the presence of morphine-resistant pain. Anesth Analg. 2003 Mar;96(3):789-795. doi: 10.1213/01.ANE.0000048088.17761.B4. PMID 12598264